CLINICAL TRIAL: NCT00150371
Title: A Multicenter, 12 Week Treatment Single Step Titration Open-Label Study Assessing The % Of Patients Achieving Ldl-C Target With Atorvastatin Starting Doses Of 10mg, 20mg, 40mg and 80mg.
Brief Title: Canadians Achieve Cholesterol Targets Fast With Atorvastatin Stratified Titration
Acronym: CANACTFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581091
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: (D006937)
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
The objective of this study is to assess the effectiveness of an atorvastatin treatment regimen involving starting doses between 10 and 80 mg, followed by a single-step titration (except for subjects started at 80mg), if required

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 79 years old
* Triglyceride level 6.8 mmol/L at screening
* LDL-C of 5.7 mmol/L at screening

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception. The latter are defined as: abstinence, surgical sterilization, oral contraceptives for at least 3 cycles, intrauterine device, implant, depot injection, or barrier method in conjunction with contraceptive foam or jelly.
* Subjects whose blood cholesterol levels are controlled (LDL-C targets) with statins other than atorvastatin
* Subjects receiving statin doses higher than the following: 10-40mg for simvastatin , 20-40mg for fluvastatin, pravastatin and lovastatin and 10-20 mg for rosuvastatin. Subjects already treated with atorvastatin at the time of screening are not eligible unless atorvastatin has been discontinued at least 2 months prior to screening
* Subjects receiving 2 or more lipid lowering agents are excluded (statins + resins or fibrates or niacin or fish oils)

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2004-06; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of subjects achieving their LDL-C target after 12 weeks of treatment according to their 10-year CHD risk category (based on the new canadian guidelines on the management and treatment of dyslipidemia).

SECONDARY OUTCOMES:
The global proportion (%) of patients reaching targets when risk categories are combined The proportion (%) of subjects achieving BOTH their LDL-C and TC/HDL-C ratio targets after 6 and 12 weeks of treatment, globally and according to their 10-year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (58):
- Canada (58):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Rothesay, New Brunswick
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Halifax, B3K 5R3, Nova Scotia
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Courtice, Ontario
  - Pfizer Investigational Site, Downsview, Ontario
  - Pfizer Investigational Site, Fort Erie, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Lindsay, Ontario
  - Pfizer Investigational Site, Markham, Ontario
  - Pfizer Investigational Site, Midland, Ontario
  - Pfizer Investigational Site, Napanee, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Niagara Falls, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, North York, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Saint Catherines, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Thunder Bay, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Montague, Prince Edward Island
  - Pfizer Investigational Site, Amos, Quebec
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Cowansville, Quebec
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Le Gardeur, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Plessisville, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint-Eustache, Quebec
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Salaberry Du Valleyfield, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste. Foy, Quebec
  - Pfizer Investigational Site, Vaudreuil, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
  - Pfizer Investigational Site, St. John's

REFERENCES:
- [Derived] Ur E, Langer A, Rabkin SW, Calciu CD, Leiter LA; CanACTFAST Study Investigators. Achieving cholesterol targets by individualizing starting doses of statin according to baseline low-density lipoprotein cholesterol and coronary artery disease risk category: the CANadians Achieve Cholesterol Targets Fast with Atorvastatin Stratified Titration (CanACTFAST) study. Can J Cardiol. 2010 Feb;26(2):80-6. doi: 10.1016/s0828-282x(10)70003-9. PMID 20151053